CLINICAL TRIAL: NCT02008136
Title: New Approaches in Evaluating Patients' Response to Botulinum Toxins in the Treatment of Chronic Neck Pain and Back Pain
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01769
Record Dates: First submitted 2013-11-27; First posted 2013-12-11 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Cervicalgia; Low Back Pain
Keywords: myofascial pain; muscle spasm; botulinum toxin; cervicalgia; lumbago; low back pain
MeSH Terms: conditions — Neck Pain; Low Back Pain; Spasm | interventions — Botulinum Toxins; Botulinum Toxins, Type A; rimabotulinumtoxinB

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- botulinum toxin injected (Experimental): Because this is an open label study, all subjects will receive one of two botulinum toxins based on their symptoms. Those will cervicalgia will receive Botox (botulinum toxin A) and those with lumbago or low back pain will receive Myobloc (botulinum toxin B)
  Interventions: Drug: Botulinum Toxins

INTERVENTIONS:
Drug: Botulinum Toxins — intramuscular injections
  Other Names: Botox; Myobloc

SUMMARY:
This protocol is a prospective, open label, pilot study examining the utility of three established pain questionnaires (the Visual Analogue Scale (VAS), Neck Disability Index (NDI), the Oswestry Low Back Pain Questionnaire and two novel pain scale devised by the PI) as well as their relationship to three novel quantitative tools to measure the effect of botulinum toxin injections for neck pain and back pain. The three novel methods for measuring neurotoxin effect are: muscle twitch patterns using surface electromyography (sEMG), cervical and lumbar range of motion using a neck and low back inclinometer, and skin surface temperature readings using an infrared imaging camera.

DETAILED DESCRIPTION:
Botulinum toxins are a well-established group of neurotoxins that have a wide variety of FDA approved clinical uses including muscle relaxation, headache prevention and bladder control. Despite the abundance of anecdotal evidence supporting their use in pain management, double blind placebo control studies examining the efficacy of botulinum toxins in the treatment of chronic neck and back pain have reported mixed findings. Several smaller studies have shown significantly positive outcomes while other studies have found no efficacy of neurotoxins compared to placebo. The existing literature reveals that most negative outcome studies were based on the Visual Analogue Scale, which is a purely subjective measure. We propose a more objective set of measures that might better reflect patients' deficits and levels of discomfort.

Our proposal is a prospective, open-label, pilot study that will examine chronic neck and back pain among veterans. Our primary specific aim is to test three novel methods for evaluating clinical deficits in patients who have chronic neck and back pain: electromyographical (EMG) activity (primary outcome) and cervical/lumbar range of motion (CROM & LROM) (primary outcome) as well as skin surface temperature (thermography) (secondary outcome). Our hypothesis is that most patients with chronic neck and back pain significantly from sustained muscle spasms. As a result, patients may exhibit surplus EMG activity in affected areas due to spontaneous muscle twitch. And consequently, they may show signs of decreased range of motion due to increased muscle tone. They may also experience a rise in skin surface temperature due to excess heat production from sustained muscle contraction. We will measure these three phenomena using three different biophysical measurement tools. Electromyographic data will be collected with a surface EMG device, and cervical and lumbar range of motion with a gravity inclinometer. Skin surface temperature will be assessed with a medical grade digital thermography camera.

The second specific aim of this study is to examine the efficacy of botulinum toxins in reversing the anomalies in the above measured parameters: to reduce excessive electromyographic activity, to increase range of motion in cervical and lumbar joints and to reduce elevated skin surface temperature. We will measure outcomes of 60 study subjects (30 for neck pain and 30 for low back pain) who will all be treated once with botulinum toxins and then followed up at 1 month, 2 months and 3 months. We will also correlate our findings with the more commonly used pain and function scales: the Visual Analogue Scale, Neck Disability Index and the Oswestry Low Back Pain Scale.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with chronic neck or back pain for at least 6 months.
* No botulinum toxin injections in the last 6 months.

Exclusion Criteria:

* Non-muscular neck or back pain
* Signs or symptoms of nerve root or spinal cord injury
* History of adverse events associated with botulinum toxin injections
* Major neurological disorder

  * recent stroke
  * myasthenia gravis
  * muscular dystrophy
  * myotonic dystrophy
  * amyotrophic lateral sclerosis
* Unstable cardiac or pulmonary disease
* Pregnancy
* Severe psychiatric illness, dementia or delirium
* Excessive obesity
* Severe spinal curvature (i.e. severe scoliosis or severe kyphosis)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Lumbar Pain Rating Scale | 3 months
  This is an 8 point rating scale for low back pain

SECONDARY OUTCOMES:
digital thermography | 3 months
  measurement of heat production from discrete muscle groups in the neck and low back using a medical grade infrared thermography camera
VAS score | 3 months
  Visual analogue scale
Oswestry Lumbar Disability Scale | 3 months
  A scoring system that assesses functional loss due to neck injury
Cervical and Lumbar Range of Motion | 3 months
  Measurement of spine rotation in x, y and z axes
surface EMG (sEMG) | 3 months
  non-invasive electrophysiological measurement of spontaneous muscle activity

CONTACTS AND LOCATIONS:
Overall Officials: Hajime A Tokuno, MD, Principal Investigator — VA Connecticut
Locations (1):
- VA Connecticut Healthcare Services, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No